CLINICAL TRIAL: NCT02013973
Title: Predictive Value of AMH (AMH=Anti Müllerian Hormone ) in IVF (IVF=In Vitro Fertilization ); a Prospective Randomized Controlled Trial
Brief Title: Predictive Value of AMH in IVF; a Prospective RCT
Acronym: AMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann Thurin Kjellberg (Other)
Responsible Party: Sponsor-Investigator, Ann Thurin Kjellberg, MD PhD, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMH Sahlgrenska
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: Anti mullerian hormone; In vitro fertilization; Optimal treatment; Randomized controlled trial
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMH-group (Experimental): The patients randomized to the AMH-group calculation of gonadotropin starting dose will be made from an algorithm including age, BMI, AFC and AMH-analysis.
  Interventions: Other: AMH-analysis
- Non-AMH-group (No Intervention): The patients randomized to the non-AMH-group, calculation of gonadotropin starting dose will be made from an algorithm including only age, BMI and AFC

INTERVENTIONS:
Other: AMH-analysis — At the first visit to the IVF-clinic a blood sample for serum-AMH is taken and frozen for later analysis in the AMH-group. The AMH assay used is the Beckman Coulter AMH Gene II assay. The analysis result will be added to the algorthm deciding what starting gonadotropin dose the patient is having.
  Arms: AMH-group

SUMMARY:
The primary aim of this trial is to compare two groups of women undergoing IVF (IVF=in vitro fertilisation ) treatment, to investigate if assessment of AMH (AMH=Anti-Müllerian hormone ), in addition to assessment of maternal age, AFC (AFC=antral follicle count ) and BMI (BMI=body mass index ) gives a more optimal COH (COH=controlled ovarian stimulation than does assessment of only age, AFC and BMI, measured as number of patients obtaining 5-12 oocytes during COH.

DETAILED DESCRIPTION:
At the first visit to the IVF-clinic a CRF (CRF=Case Report Form) of demographics will be filled in regarding age, BMI, parity, presence of PCOS (PCOS=polycystic ovarian syndrome ), smoking and duration of infertility and a blood sample for serum-AMH is taken and frozen for later analysis. The serum-AMH level is constant during the menstrual period (La Marca et al 2006) and a blood sample can be taken on any cycle day. The AMH assay used is the Beckman Coulter AMH Gene II assay. Classification of the serum AMH values into expected low-, normal-, or high ovarian response is based on the data presented a large prospective cohort study of patients going through COH (Nelson et al 2009). Since that publication used an older assay the reference intervals are calculated and translated as described in a recent publication on AMH assays (Nelson et al 2012). Serum-AMH level increases during GnRH (GnRH= gonadotropin releasing hormone) agonist downregulation (Jayaprakasan et al 2008), thus the blood sample is preferably taken before start of down-regulation. A long GnRH agonist treatment protocol is used. Patients are down-regulated with GnRH agonist from luteal phase, or first cycle day when anovulatory patient, until estradiol is < 200 pmol/l. After down-regulation, an assessment of AFC will be performed by sonography, and the patient will be randomized.

For the patients randomized to the AMH-group calculation of gonadotropin starting dose will be made from an algorithm including age, BMI, AFC and serum-AMH. For the patients randomized to the non-AMH-group, calculation of gonadotropin starting dose will be made from an algorithm including only age, BMI and AFC. The AMH blood sample in this group will be analyzed after completion of the study.

Stimulation is started with a dose of rFSH (rFSH=recombinat follicle stimulating hormone) calculated according to the dose algorithms used in the two groups. The name of the gonadotropin preparation, the dose and number of treatment days will be recorded. The same applies for all drugs used. Monitoring will be performed with mandatory estradiol on the day of stimulation start and on stimulation day 6. The dose of gonodotropin can be adjusted on day 7. If estradiol is > 1200 pmol/l the dose is reduced with one step according to the dose algorithm. If estradiol is < 350 pmol/l the dose is increased with one step according to the dose algorithm. Vaginal sonography is performed on stimulation day 9-11 to estimate the number and size of follicles. The number of follicles >10 mm at sonography 0-2 days before ovulation induction is recorded. Ovulation induction with 6500 IU (IU=international units) rHCG (rHCG=recombinant human chorion gonadotropin ) is given when >=2 follicles >=17 mm. 36 hours after ovulation induction transvaginal oocyte pickup is performed according to standard procedure at the clinic using sedation and paracervical administration of local anaesthetics, and all follicles > 10 mm are punctured. The oocytes will be fertilized using standard IVF procedure. In the case of an unexpected poor semen sample on the day of ovum pick-up microinjection will be performed. The fertilization rate is recorded. Embryo transfer is done on day 2 or 3 according to routine procedures in the clinic. In the case of no GQE (GQE=good quality embryos ) it is allowed to perform double embryo transfer, otherwise single embryo transfer is mandatory. Luteal phase support using vaginal route is given from the day of embryo transfer and for 14 more days, until pregnancy test (urinary ). In case of impending OHSS (OHSS=ovarian hyperstimulation syndrome ), where decision is made to cryopreserve all embryos, the outcome of the first transfer of a cryopreserved embryo will be included in the study results for secondary endpoints. In case of pregnancy, an early vaginal sonography is performed in pregnancy week 7-8. The number of cancelled cycles due to poor response is recorded. The number of patients having moderate or severe OHSS, requiring intervention, will be recorded until four weeks after ovum pick up.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for IVF with standard method for the couple exists (i.e. more than one year of infertility and work-up has been performed suggesting IVF as the proper treatment and no known severe male factor exists).
2. Age >18 and < 40 years.
3. BMI > 18 and < 35.
4. First IVF treatment for the woman.
5. Willing to participate in randomization between intervention group and control group and to sign informed consent.

   -

Exclusion Criteria:

1. IVF with ICSI (ICSI=intracytoplasmic sperm injection ) planned.
2. Oocyte donation planned.
3. Treatment with PGD (PGD=preimplantation genetic diagnosis ) planned.
4. Medical or psychological condition indicating ineligibility for the study.
5. Patient with insufficient knowledge of Swedish language to understand patient information.
6. Previous participation in this study.

   -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients obtaining 5-12 oocytes during COH | 2 years

SECONDARY OUTCOMES:
Cancelled cycle rate | 2 years
Total dose of gonadotropins | 2 years
Number of participants developing moderate or severe OHSS | 2 years
  Follow-up of OHSS rate performed 4 weeks after ovum pick up
Embryology | 2 years
  Number of oocytes retrieved, fertilization rate, number of good quality embryos, number of surplus embryos possible to cryopreserve, number of embryos transferred
Pregnancy and live birth rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christina Bergh, MD PhD, Study Chair — Sahlgrenska University Hospital; Ann Thurin-Kjellberg, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Reproductive medicine,, Gothenburg, Sweden

REFERENCES:
- [Derived] Magnusson A, Olerod G, Thurin-Kjellberg A, Bergh C. The correlation between AMH assays differs depending on actual AMH levels. Hum Reprod Open. 2017 Dec 8;2017(4):hox026. doi: 10.1093/hropen/hox026. eCollection 2017. PMID 30895238